# **SUMMARY OF CHANGES**

NCI Protocol #: 10411 Local Protocol #: 21-070

Protocol Version Date: April 4, 2025

**Protocol Title:** Phase 2 Study of Rogaratinib (BAY 1163877) in the Treatment of Patients with Sarcoma Harboring Alterations in Fibroblast Growth Factor Receptor (FGFR) 1-4 and SDH-

deficient Gastrointestinal Stromal Tumor (GIST)

**Informed Consent Version Date:** April 4, 2025

# **SUMMARY OF CHANGES – Consent**

# I. Study team-initiated Consent Changes:

| # | Section | Comments |
|---|---|---|
| 1 | Header | Updated the protocol version date. |
| 2 | Patient Study<br>Calendar | Updated Patient Study Calendar. The reference to "Cycle 29" is an error. It should reference "Cycle 27" as the Day 1 visit when the Cycle 26 scan will be reviewed. After Cycle 27 Day 1, scans will occur every 3 cycles, so the next scan review visit will occur on Cycle 30 Day 1, Cycle 33 Day 1, etc. Also edited "Medical imaging scans for tumor measurements" to specify "through <i>the end of</i> Cycle 26, and then every 3 cycles thereafter." |

# **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the anti-cancer drug, rogaratinib (BAY 1163877), for treatment of advanced sarcoma with alteration in fibroblast growth factor receptor (FGFR 1-4), and in patients with SDH-deficient gastrointestinal stromal tumor (GIST).

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: P10411, Phase 2 Study of Rogaratinib (BAY 1163877) in the Treatment of Patients with Sarcoma Harboring Alterations in Fibroblast Growth Factor Receptor (FGFR) 1-4 and SDH-deficient Gastrointestinal Stromal Tumor (GIST) (NCT# NCT04595747)

# **Overview and Key Information**

# What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have sarcoma, and your cancer has a change in a group of proteins called the FGFRs (fibroblast growth factor receptors), or you have a type of sarcoma called SDH-deficient GIST (succinate dehydrogenase deficient gastrointestinal stromal tumor).

# Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

This study is being done to answer the following question:

Can we lower the chance of your sarcoma growing or spreading when treated with the anticancer drug rogaratinib (BAY 1163877)?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your sarcoma. The usual approach is defined as care most people get for sarcoma.

# What is the usual approach to my sarcoma?

The usual approach for patients with sarcoma with an FGFR alteration who are not in a study is treatment with chemotherapy using one of the following: doxorubicin, ifosfamide, trabectedin, dacarbazine, platinum compounds, doxorubicin plus ifosfamide, doxorubicin plus ifosfamide and dacarbazine, pazopanib, or gemcitabine with docetaxel, vinorelbine or dacarbazine. Patients with SDH-deficient GIST may be treated with imatinib, sunitinib or regorafenib. These drugs are approved by the Food and Drug Administration (FDA). There are no treatments that are proven to cure patients with your type of cancer.

# What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

# What will happen if I decide to take part in this study?

If you decide to take part in this study, you will receive rogaratinib (BAY 1163877) for as long as this treatment is helping you and not causing side effects that are too severe.

After you finish your treatment, your doctor will continue to follow your condition and watch you for side effects for an additional 30 days. Your doctor will call you on the phone approximately 30 days after your last dose of study drug to evaluate any remaining symptoms.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the study drug may not be as good as the usual approach for your cancer at shrinking or stabilizing your cancer.

There is also a risk that you could have side effects from the study drug. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Diarrhea
- Tiredness
- Loss of appetite

There may be some risks that the study doctors do not yet know about.

### **Benefits**

This drug has shrunk your type of cancer in animals or in living human or living animal cells. It is unlikely that it will work in everyone with your cancer or help you live longer. This study may help the study doctors learn things that may help other people in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

# Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (National Cancer Institute [NCI]). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

# What is the purpose of this study?

The purpose of this study is to test the good and bad effects of the investigational study drug called rogaratinib (BAY 1163877). Investigational means that the study drug, Rogaratinib (BAY

1163877), is not approved by the FDA for your type of cancer. Rogaratinib (BAY 1163877) could shrink your cancer, but it could also cause side effects, which are described in the risks section below. The study doctors hope to learn if the study drug will shrink the cancer.

We don't know if rogaratinib (BAY 1163877) works to treat cancer in people, but it has shrunk several types of tumors in animals. Rogaritinib (BAY 1163877) has also been given to some people with other types of cancer.

There will be about 48 people taking part in this study.

# What are the study groups?

For patients who do not have SDH-deficient GIST, this study has a screening step. The purpose of this step is to review information about your tumor using the results of tests you have had done on your tumor prior to this study to find out if it has a specific change in proteins called fibroblast growth factor receptors (FGFRs). If your tumor has an FGFR alteration and you meet all the study requirements, then we can assign you to the study based on these changes. If we find that your tumor does not have the changes in FGFRs that are needed for this study, then your doctor will discuss other options for your care. Patients with SDH-deficient GIST do not require this screening test.

In this study, all participants will receive the study drug rogaratinib (BAY 1163877).

Dosing schedule: You will take rogaratinib (BAY 1163877) tablets by mouth, twice a day, every day of each cycle. You should take the rogaratinib (BAY 1163877) with 8 oz of water. It can be taken with or without food. Rogaratinib (BAY 1163877) tablets should be swallowed whole. Do not chew. On Day 1 of Cycles 1-3 and Day 15 of Cycle 1 and 2, you will bring your morning dose of rogaratinib (BAY 1163877) with you to the clinic. Each cycle lasts 28 days. See the study calendar for more information.

You will not be able to get additional doses of the drug.

# What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if you are eligible to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

These exams, tests, and procedures to monitor your safety and health include:

• An eye exam before you begin the study.

This study will use genetic tests that may identify changes in the genes in your DNA. Your genes carry information about you and your family, from the color of your eyes to health conditions for which you may be at risk, such as certain kinds of cancer.

Finding these changes would not affect your treatment in this study. However, they could affect your health in other ways. You and your doctor will not receive the results of these tests.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

You will be asked to have biopsies for the study and we will also request that a portion of your tumor that was previously removed and stored in a pathology archive (archival tissue), if available, be sent to a central laboratory. The study biopsy takes small pieces of cancer tissue from your body. This is like the biopsy you had that helped diagnose your cancer. The first biopsy will be done before you begin the study drug. This biopsy and the archival tissue is being collected to evaluate whether the genetic changes in the tumor in FGFR and related proteins are still present immediately prior to starting on study. This biopsy and the archival tissue will also allow us to evaluate the genes in your tumor and evaluate if this is related to response to rogaratinib (BAY 1163877). However, a biopsy may not be collected if your doctor thinks that a biopsy is not safe and has discussed this with the Study Chair. A second optional biopsy will be done if your disease gets worse.

Blood samples will also be taken for the study. Blood sample will be collected before you begin the study treatment, before you take rogaratinib (BAY 1163877) on the days you visit the clinic on cycle 1 day 15, cycle 2 day 1, cycle 2 day 15, cycle 3 day 1, and on the day you visit the clinic if you need to have your dose of rogaratinib (BAY 1163877) lowered.

Researchers will obtain genetic material (DNA and RNA) from your tumor tissue and blood samples. Your tumor DNA and RNA will be sequenced to evaluate changes in your tumor DNA and RNA that may occur during treatment. You and your study doctor will not get any results of this testing. If you agree to take part in the study, you may need to sign a separate consent form for the study biopsy at the hospital or clinic where the biopsy is done.

A patient study calendar is attached at the end of this document. It shows how often these procedures will be done.

# What risks can I expect from taking part in this study?

### **General Risks**

If you choose to take part in this study, there is a risk that the study drug may not be as good as the usual approach for your cancer at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The drug used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 4 months after you have completed the study.

# **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection, significant bleeding, or collapsing of the lung can occur. You may sign a separate consent form for the study biopsy that describes the risks in more detail.

### **Blood Draw Risks**

Some of the risks from drawing blood from your arm may include pain, bruising, light-headedness, and rarely, infection. For most people, needle punctures to get blood samples do not cause any serious harm. Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

# **Side Effect Risks**

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drugs.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

You should notify your doctor immediately at the first sign of poorly formed or loose stools or an increased frequency of bowel movements. Loperamide (Imodium) should be kept on hand and should be taken as recommended by your doctor.

# **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

### Risk Profile for Rogaratinib (BAY 1163877)

(Table Version Date, February 14, 2023)

### COMMON, SOME MAY BE SERIOUS

In 100 people receiving rogaratinib (BAY 1163877), more than 20 and up to 100 may have:

- Diarrhea
- Tiredness
- Loss of appetite
- Hair loss

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving rogaratinib (BAY 1163877), from 4 to 20 may have:

- Visual loss
- Dry mouth, skin
- Sores in the mouth which may cause difficulty swallowing
- Nausea, vomiting
- Pain in joints
- Changes in taste
- Change in or loss of some or all of the finger or toenails
- Nail ridges

# **Additional Drug Risks**

Rogaratinib can cause increased levels of phosphorous in your blood. This will be monitored and is a common side effect. If this happens, it may require you to take medications to lower phosphorous, reduce the amount of phosphorous in your diet, interrupt drug dosing, or have the dose reduced.

The study drug could interact with other drugs and food especially certain immunosuppressants anesthetics, antipsychotics, certain drugs used to treat migraine headache, and grapefruit juice, which can alter the drug levels in your blood. Ask your study doctor before starting any new medications. Your study doctor will give you a drug information handout and wallet card that lists these possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

# What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take the study drug at home.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby or donate sperm while taking part in this study. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 4 months after your last dose of study drug.

For women of childbearing potential and men: You must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before you begin the study, for the duration of study participation, and 4 months after completion of your last dose of the study drug.

# What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the costs of getting rogaratinib (BAY 1163877) ready and giving it to you.
- the eye exams conducted before you begin your study.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

- The biopsy to confirm changes in the group of proteins called FGFRs and to test your response to treatment, before you begin the study and when your disease gets worse.
- The archival tumor sample collection to evaluate the genes in your tumor and evaluate if this is related to response to rogaratinib (BAY 1163877).
- The blood collection to evaluate your response to treatment before you begin the study.
- The blood collection to evaluate the level of rogaratinib (BAY 1163877) before you begin the study treatment, before you take rogaratinib (BAY 1163877) on the days you visit the clinic (e.g., cycle 1 day 15, cycle 2 day 1, cycle 2 day 15, cycle 3 day 1, etc.), and on the day you visit the clinic if you need to have your dose of rogaratinib (BAY 1163877) lowered.

You or your insurance provider will not have to pay for the rogaratinib (BAY 1163877) while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

# Some of these organizations are:

- The study sponsor and any company supporting the study now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study

doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

# Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

# Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for, but cannot complete any of these studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

# Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or

straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

### **Known future studies**

If you choose to take part in this optional study, researchers will collect your blood to evaluate the level of Rogaratinib (BAY 1163877) and tumor tissue for research on evaluating the changes in your DNA and RNA that occur during treatment. Researchers will obtain genetic material (DNA and RNA) from your tumor cells. Your DNA and RNA will be used for genomic sequencing, which is sequencing of all or part of your DNA. All your genetic information makes up your genome. Genomic sequencing is a test that records all or part of the pieces of DNA that are in your genes, piece by piece. This is usually done to look for changes in your genome that may cause health problems. The genomic sequencing will be done by an NCI-supported laboratory in Frederick, Maryland, known as the National Clinical Laboratory Network (NCLN) Genomics Laboratory at the Frederick National Laboratory for Cancer Research. The laboratory will compare the genomic sequences from your tumor and blood cells to identify how they differ. The differences between genomic sequences of your tumor and blood cells may be important to understand why you did or did not respond to the treatment you received. Researchers hope to find potential "biomarkers" (changes present in tumor tissue that predict how patients with your type of cancer may respond to current or future treatments). This optional study may improve the ability to select future treatments or treatment combinations for others in the future. This optional study will not affect the cancer treatment or approach that you receive.

Neither you nor your study doctor will be informed when the genetic sequencing research will be done. You and your study doctor will not receive reports of these studies, as they are intended for research purposes only and cannot be used to plan treatment.

### Unknown future studies

If you choose to take part in this optional study, any of your tumor tissue or blood samples left over from the genomic sequencing will be stored. Storing samples for future studies is called "biobanking." The biobank is being run by the Nationwide Children's Hospital in Columbus, Ohio, and is supported by the NCI. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we do not know what research may be done in the future using your tumor tissue and blood samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.

- Future research studies may include genomic sequencing.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes. If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

# What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. A sample of tissue will be collected from an optional extra biopsy if your disease gets worse. For the biopsy procedure, the study doctor will use a needle to take pieces of your tumor. This process may be repeated several times in the same appointment in order to get enough tissue. About 1 teaspoon of blood will be collected from a vein in your arm if your disease gets worse.
- 2. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 3. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 4. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

# What are the risks in this optional sample collection?

- The most common risks related to a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection, significant bleeding, or collapsing of the lung can occur. The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone outside of the research study could get access to your study records or trace information in a database back to you. They could use that information in a way that could harm you. Researchers believe the chance that someone could access and misuse your information is

- very small. However, the risk may increase in the future as people find new ways of tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: <a href="https://www.genome.gov/10002328/">https://www.genome.gov/10002328/</a>

# How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information. Only your study doctor and a few study researchers will have access to the master list linking the code numbers to names. The biobank and the genomic sequencing laboratory will receive your samples with the following information only: your sample code number; your age, race/ethnicity, and sex; your type of cancer; any previous treatments you received for your cancer; and the treatment you will receive for this current study.
- 2. Researchers who study your samples and information will not know who you are. They also must agree that they will not try to find out who you are. The researchers must be trained in the handling of private information. Any researcher who wants to study your stored samples and genetic information must apply and be approved to do so.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance for exams, tests, and procedures done for research purposes only; these include the biopsy, blood draw, DNA/RNA sequencing, and biobanking of your specimen(s). You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What if I change my mind about this optional sample collection?

If you decide you no longer want your samples to be used, you can call the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main

trial\*), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

### What if I need my tissue or blood samples to be returned?

Tumor tissue or blood samples that remain in the biobank can be returned if needed for medically necessary events or procedures to assure appropriate medical care, such as for DNA or RNA analysis. Specimens may also be returned if tissue is needed to determine eligibility for enrollment in a research protocol or clinical trial. Every effort will be made to facilitate medically necessary events or procedures to assure appropriate medical care for a patient with a serious or lifethreatening illness.

Tumor tissue or blood samples and genetic material (DNA and RNA) that is no longer in the biobank or that has already been given to or used by researchers cannot be returned. No samples will be returned for matters related to patients needing or wanting genetic testing to determine medically important risks.

# What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*).

Please circle your answer below to show if you would or would not like to take part in each optional study:

### Samples for known future studies:

I agree that my samples and related health information may be used for the laboratory or studies described above.

YES NO

### Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

### Contact for Future Research

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

This is the end of the section about optional studies.

# My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

# Participant's signature

Date of signature

# Signature of person(s) conducting the informed consent discussion

Date of signature

Protocol Version Date 04/04/2025

10411 Page 19 of 18

# Patient Study Calendar

| | Before you | | Cycle | Cycles 1 - 4 | | Cycles 5 - 26 | Cycle 27 and Every 3 Cycles Thereafter | After you finish the study treatment |
|---|---|---|---|---|---|---|---|---|
| | study | Day 1 | Day 8 | Day 15 | Day 22 | Day 1 | Day 1 | |
| Rogaratinib (BAY 1163877)^ | | X | | | | | Χ | |
| Pre-study procedures including Informed consent,<br>Demographics, Medical history, and Weight | × | | | | | | | |
| Concurrent meds | × | | × | | | | Χ | × |
| Physical exam and Vital signs | × | × | | × | | × | × | × |
| An assessment of how you perform everyday activities and tasks | × | | | | | | | |
| Blood draws for complete blood count | × | × | | × | | × | × | × |
| Blood draws to evaluate your general health status | × | × | | × | | × | × | × |
| Side effects evaluation | | | Χ | | | | X | × |
| Medical imaging scans for tumor measurements | X <sup>B</sup> | Scans are | done ever<br>thei | /8 weeks tl | very 8 weeks through the end<br>then every 3 cycles thereafter | Scans are done every 8 weeks through the end of Cycle 26, and then every 3 cycles thereafter | × | × |
| Pregnancy test (for women of child-bearing potential only) | × | | | | | | | |
| Eye exam | Xc | | | | | | | |
| ECG (as your doctor indicates it is needed) | × | | | | | | | |
| Archival tissue (if available) | × | | | | | | | |
| Mandatory tumor tissue collection for research purposes | Xc | | | | | | | |
| Optional tumor tissue collection for research purposes | | | | | | | | × |
| Blood Collection for research purposes | × | | | | | | | |
| Blood Collection to evaluate the level of<br>Rogaratinib (BAY 1163877) <sup>D</sup> | × | × | | × | | | | |

# Protocol Version Date 04/04/2025

| $\overline{}$ | $\infty$ |
|---------------|----------|
| 4 | f 1 |
| Ò | 0 |
| _ | 20 |
| | e |
| | O |
| | Ра |

| | | Before you | | Cycle | Cycles 1 - 4 | | Cycles 5 - 26 | Cycle 27 and Every 3 Cycles Thereafter | After you finish the study treatment |
|---|---|---|---|---|---|---|---|---|---|
| | | study | Day 1 | Day 8 | Day 15 | Day 22 | Day 1 | Day 1 | |
| Optional Blood Collection to evaluate the level of Rogaratinib (BAY 1163877) | aluate the level of | | | | | | | | × |
| | A: Rogaratini | b (BAY 1163877) do | ose as assig | ned. Take t | twice a day | with 8 oz wa | ter, with or without | A: Rogaratinib (BAY 1163877) dose as assigned. Take twice a day with 8 oz water, with or without any moderate fat or low fat diet. Swallow whole. Do not chew. | e. Do not chew. |
| | B: Imaging su | ch as scans or X-ra | ys will be d | one within | 4 weeks be | fore you begi | B: Imaging such as scans or X-rays will be done within 4 weeks before you begin study treatment. | | |
| | C: May be do<br>required a | May be done ≤ 14 days before you begin study<br>equired after discussion with the Study Chair. | e you begir<br>η the Study | ו study trea<br>Chair. | tment. A bi | opsy will be c | collected if deemed s | May be done ≤14 days before you begin study treatment. A biopsy will be collected if deemed safe by your doctor. If your doctor thinks that a biopsy is not safe, a biopsy may not be required after discussion with the Study Chair. | olopsy is not safe, a biopsy may not be |
| | D: Blood colle<br>1, cycle 2 o | Blood collection will be performed before you be<br>1, cycle 2 day 15, cycle 3 day 1, etc.), and on the | rmed befor<br>1, etc.), anc | re you begir<br>I on the day | the study<br>/s you visit 1 | treatment, bι<br>the clinic afte | egin the study treatment, before you take rogara<br>days you visit the clinic after a dose reduction. | Blood collection will be performed before you begin the study treatment, before you take rogaratinib (BAY 1163877) on the days you visit the clinic (e.g., cycle 1 day 15, cycle 2 day 15, cycle 3 day 1, etc.), and on the days you visit the clinic after a dose reduction. | inic (e.g., cycle 1 day 15, cycle 2 day |